CLINICAL TRIAL: NCT00497965
Title: Pilot Study: Does Chiropractic Care Decrease Fall Risk in Older Adults?
Brief Title: Pilot Study: Does Chiropractic Care Decrease Fall Risk in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Chiropractic College (Other)
Collaborators: Foundation for Chiropractic Education and Research (FCER) (Other)
Responsible Party: Dr. Cheryl Hawk, Cleveland Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-07252006; FCER 06-10-02
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Musculoskeletal Equilibrium
Keywords: Balance; Chiropractic; Older Adults
MeSH Terms: interventions — Manipulation, Chiropractic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Chiropractic Manipulation
Behavioral: Balance Exercises

SUMMARY:
The purpose is to study the effect of chiropractic care on balance in older adults.

DETAILED DESCRIPTION:
The specific aims of this pilot study are to: 1) build a recruitment pool of older adults within the local community; 2) establish a protocol for long-term surveillance of falls for older adult chiropractic patients; 3) explore dose-response patterns to chiropractic care by comparing Berg Balance Scale scores at 12 months from baseline in three groups of older adults with impaired balance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 or older
2. Able to stand steadily without assistance on one leg for an average of <5 seconds (determined by averaging the time for both legs)
3. Able to attend all scheduled sessions (by self-report)

Exclusion Criteria:

1. Non-ambulatory (wheelchair-bound); this precludes required balance testing; however, volunteers requiring assistive devices such as canes and walkers are not excluded
2. received chiropractic care or other manual care within the past three months (by self-report)
3. initiated exercise program for balance / lower body strength within the past month (by self-report)
4. contraindications to SMT or mild-exertion exercise, as determined by the clinician through physical exam and x-rays (if indicated). Contraindications include but are not limited to: signs and symptoms associated with vertebrobasilar insufficiency (including facial numbness, diplopia, drop attacks, dysphagia, and ataxia which are not fatiguable or habituable with repeated provocative head positioning); unstable or severe medical condition; severe osteoporosis, fracture or other osseous abnormalities; "high cardiovascular risk", i.e. persons with known severe cardiovascular, pulmonary or metabolic disease, or one or more major signs/symptoms suggestive of cardiovascular and pulmonary disease
5. absence of indications for SMT, as determined by the clinician through history, physical exam, orthopedic tests, and static and motion palpation. Indications for SMT include identification of decreased or increased spinal joint mobility usually accompanied by tenderness and muscle tension and spasm;
6. unable to understand English adequately to complete study forms and questionnaires, because we do not have study personnel fluent in other languages;
7. central causes of vertigo, including arteriovenous malformations, cerebral hemorrhage, brainstem vascular disease, tumors and demyelenating diseases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mean change scores for the BBS from baseline to 8 weeks will be compared with a one-factor analysis of variance. Post-hoc comparisons of means and associated confidence intervals will be evaluated using the Tukey test. | Through December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Hawk, D.C., Ph.D., Principal Investigator — Cleveland Chiropractic College
Locations (1):
- Cleveland Chiropractic College Health Center, Kansas City, Missouri, United States